CLINICAL TRIAL: NCT01610206
Title: A Randomized Open Label Phase II Study of Weekly Gemcitabine Plus Pazopanib Versus Weekly Gemcitabine Alone in the Treatment of Patients With Persistent or Relapsed Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma
Brief Title: A Randomized Study of Safety and Efficacy of Pazopanib and Gemcitabine in Persistent or Relapsed Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Linda R Duska (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Linda R Duska, Associate Professor, Division of Gynecology Oncology, University of Virginia, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16153
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Results first posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: recurrent; persistent
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Recurrence | interventions — Gemcitabine; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gemcitabine (Active Comparator)
  Interventions: Drug: Gemcitabine
- Gemcitabine + pazopanib (Experimental)
  Interventions: Drug: Gemcitabine; Drug: pazopanib

INTERVENTIONS:
Drug: Gemcitabine — Patients will receive gemcitabine 1000 mg/m2 administered weekly on days 1 and 8 (30 minutes IV infusion) of each cycle for up to 6 cycles. Each cycle is 21 days.
  Other Names: gemzar
Drug: pazopanib — Patients will receive pazopanib 800mg PO daily on days 1-21 of treatment cycles
  Other Names: votrient
  Arms: Gemcitabine + pazopanib

SUMMARY:
Ovarian cancer is the leading cause of gynecologic cancer deaths, and the fifth most common cause of cancer deaths in women. While approximately 75% of patients with epithelial ovarian cancer will respond to first-line chemotherapy with platinum and paclitaxel, most patients with advanced stage epithelial ovarian cancer will experience disease recurrence. Pazopanib is a novel agent has recently been approved for the treatment of subjects with advanced renal cell carcinoma (RCC), and preclinical studies suggest it may be effective in other cancers such as ovarian cancer. Therefore, the purpose of this study is to test the efficacy and safety of a novel agent, pazopanib, as an adjunct to a standard treatment, gemcitabine, for recurrent or persistent ovarian cancer. This is an open label study in which subjects will be randomized 1:1 to receive 4 cycles of either gemcitabine, or gemcitabine with pazopanib. Gemcitabine will be administered as an IV infusion weekly on days 1 and 8 of a 21 day cycle. Subjects randomized to receive pazopanib will take 800 mg daily during the 21 day cycle. All subjects will be monitored for toxicity and other indicators of safety (labs, physical exams, vitals) at intervals throughout the treatment cycles. Subjects will be followed for up to 5 years following the conclusion of treatment to evaluate efficacy. The primary endpoints of the study are progression free survival and overall survival, which will be assessed at three years.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old
* Must have measurable or detectable ovarian, fallopian or primary peritoneal cancer
* Must have been treated previously with carboplatin, cisplatin or another organoplatinum compound

Exclusion Criteria:

* Women who are pregnant or nursing
* History of congenital long QT syndrome
* Active bleeding or at risk of a bleeding disorder
* Other significant medical condition or history of medical condition which may put the patient at risk

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Duska, MD, Study Director — University of Virginia School of Medicine
Locations (8):
- United States (8):
  - Maine Medical Center (MMP Women's Health), Scarborough, Maine
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Duke University, Durham, North Carolina
  - Stephenson Cancer Center University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - MD Anderson, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Wisconsin-Madison, Madison, Wisconsin

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Duska LR, Petroni GR, Varhegyi N, Brown J, Jelovac D, Moore KN, McGuire WP, Darus C, Barroilhet LM, Secord AA. A randomized phase II evaluation of weekly gemcitabine plus pazopanib versus weekly gemcitabine alone in the treatment of persistent or recurrent epithelial ovarian, fallopian tube or primary peritoneal carcinoma. Gynecol Oncol. 2020 Jun;157(3):585-592. doi: 10.1016/j.ygyno.2019.10.014. Epub 2020 Apr 1. PMID 32247603

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine | Gemcitabine + Pazopanib
Started | 73 | 75
Completed | 63 | 45
Not Completed | 10 | 30
Not completed — Adverse Event | 10 | 30

BASELINE CHARACTERISTICS:
Population: All eligible and randomized participants who received study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine | Gemcitabine + Pazopanib | Total
Number analyzed (Participants) | 73 | 75 | 148
Age, Continuous [Mean (Full Range); unit: years] | 62 [38 to 82] | 63 [30 to 80] | 63 [30 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 75 | 148
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 8 | 12
  White | 58 | 57 | 115
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 73 | 75 | 148

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-Free Survival (PFS) is defined as the duration of time from study entry to time of recurrence/progression or death from any cause, whichever occurs first.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine | Gemcitabine + Pazopanib
Number analyzed (Participants) | 73 | 75
months | 2.9 [2.1 to 4.1] | 5.3 [4.2 to 5.8]
Statistical Analysis 1: Comparison: Gemcitabine vs Gemcitabine + Pazopanib; Test type: Equivalence — To estimate the progression-free survival hazard ratio of the combination of weekly gemcitabine and pazopanib compared to weekly gemcitabine alone in patients with persistent or recurrent ovarian, fallopian tube, or primary peritoneal cancer; p = 0.019, non-parametric weighted Tarone-Ware test; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.61 to 1.07]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events will be evaluated using CTCAE criteria from the start of study treatment until 30 days following the last dose of study treatment
Time Frame: 30 days after last dose
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine | Gemcitabine + Pazopanib
Number analyzed (Participants) | 73 | 75
Participants | 73 | 75

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the first study-related procedure was performed until 30 days post administration of the last study treatment.
Arm/Group | Gemcitabine | Gemcitabine + Pazopanib
All-Cause Mortality (participants affected / at risk) | 54/73 | 63/75
Serious Adverse Events (participants affected / at risk) | 20/73 | 63/75
Other Adverse Events (participants affected / at risk) | 73/73 | 75/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine (N=73) | Gemcitabine + Pazopanib (N=75)
Anemia (Blood and lymphatic system disorders) | 2 | 8
Neutropenia (Investigations) | 15 | 30
Thrombocytopenia (Investigations) | 2 | 11
Fatigue (General disorders) | 1 | 9
Elevated AST (Investigations) | 1 | 9
Hypertension (Vascular disorders) | 1 | 12
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Fever (General disorders) | 1 | 0
ALT increased (Investigations) | 1 | 9
Decreased lymphocyte count (Investigations) | 0 | 2
White blood cell count (Investigations) | 1 | 11
Hyponatremia (Metabolism and nutrition disorders) | 0 | 5
Headache (Nervous system disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine (N=73) | Gemcitabine + Pazopanib (N=75)
anemia (Blood and lymphatic system disorders) | 26 | 11
febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
heart failure (Cardiac disorders) | 0 | 1
tinnitus (Ear and labyrinth disorders) | 3 | 1
vertigo (Ear and labyrinth disorders) | 0 | 2
Hypothyroidism (Endocrine disorders) | 0 | 2
blurred vision (Eye disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 7
Bloating (Gastrointestinal disorders) | 0 | 4
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 7 | 10
Diarrhea (Gastrointestinal disorders) | 7 | 24
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Fecal incontinence (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 2
Gastroesophageal reflux (Gastrointestinal disorders) | 1 | 5
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 2
Gastroparesis (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 4 | 13
Nausea (Gastrointestinal disorders) | 18 | 35
Oral pain (Gastrointestinal disorders) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 5 | 19
Chills (General disorders) | 4 | 6
Edema face (General disorders) | 0 | 1
Edema limbs (General disorders) | 4 | 5
Fatigue (General disorders) | 28 | 41
Fever (General disorders) | 4 | 4
Flu-like symptoms (General disorders) | 3 | 4
Gait disturbance (General disorders) | 0 | 1
Infusion related reaction (General disorders) | 1 | 0
Injection site reaction (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Pain (General disorders) | 1 | 2
Mucosal infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 2
Alanine Aminotransferase increased (Investigations) | 5 | 15
Alkaline Phosphatase increased (Investigations) | 3 | 12
Aspartate Aminotransferase increased (Investigations) | 5 | 22
Blood bilirubin increased (Investigations) | 0 | 2
Creatinine increased (Investigations) | 2 | 6
Neutrophil count decreased (Investigations) | 4 | 8
Platelet count decreased (Investigations) | 3 | 12
Weight loss (Investigations) | 0 | 4
White blood cell decreased (Investigations) | 3 | 14
Anorexia (Metabolism and nutrition disorders) | 9 | 21
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 5
Hypermagnesmia (Metabolism and nutrition disorders) | 0 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 2 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 7
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 5
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Extremity pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Cognitive disturbance (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 5
Dysgeusia (Nervous system disorders) | 1 | 6
Headache (Nervous system disorders) | 6 | 17
Paresthesia (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 8
Tremor (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 2
Urinary tract pain (Renal and urinary disorders) | 2 | 0
Dyspareunia (Reproductive system and breast disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Palmar-Plantar Erythrodysethesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 2
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Hot flashes (Vascular disorders) | 2 | 2
Hypertension (Vascular disorders) | 0 | 17
Hypotension (Vascular disorders) | 0 | 1
Lymphedema (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
Our study is limited by lack of placebo control, independent pathology and radiologic review, and correlative science. We did not collect data regarding quality of life, and the study was performed in an unselected patient population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Informed Consent Form (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT01610206/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-03-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT01610206/Prot_SAP_001.pdf